CLINICAL TRIAL: NCT03302897
Title: A Phase 1, Open Label, Antigen Dose-Escalation Clinical Trial to Evaluate the Safety, Tolerability, and Immunogenicity of LEP-F1 + GLA-SE in Healthy Adult Subjects
Brief Title: Phase 1 LEP-F1 + GLA-SE Vaccine Trial in Healthy Adult Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Access to Advanced Health Institute (AAHI) (Other)
Collaborators: American Leprosy Missions (Unknown)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: IDRI-LEPVPX-118
Record Dates: First submitted 2017-10-02; First posted 2017-10-05 (Actual); Last update posted 2019-04-11 (Actual); Status verified 2019-04

CONDITIONS: Leprosy
Keywords: Leprosy, vaccine, adjuvant, GLA, GLA-SE
MeSH Terms: conditions — Leprosy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- 2 μg LEP-F1 + 5 μg GLA-SE (Experimental): Three intramuscular injections of LEP-F1 + GLA-SE at Days 0, 28, and 56. Low dose of antigen.
  Interventions: Biological: LEP-F1 + GLA-SE
- 10 μg LEP-F1 + 5 μg GLA-SE (Experimental): Three intramuscular injections of LEP-F1 + GLA-SE at Days 0, 28, and 56. Higher dose of antigen.
  Interventions: Biological: LEP-F1 + GLA-SE

INTERVENTIONS:
Biological: LEP-F1 + GLA-SE — Investigational vaccine

SUMMARY:
The purpose of this study is to compare the safety, tolerability, and immunogenicity in healthy adult subjects of an investigational vaccine being developed for the prevention of leprosy. Two dose levels of the vaccine will be evaluated.

DETAILED DESCRIPTION:
The purpose of this study is to compare the safety, tolerability, and immunogenicity of the LEP-F1 + GLA-SE vaccine. The vaccine consists of the recombinant four-antigen Mycobacterium leprae antigen LEP-F1 in combination with the adjuvant formulation GLA-SE (Glucopyranosyl Lipid A - Stable Emulsion) and is being developed for the prevention of leprosy disease. This is a first-in-human study and will be conducted in healthy adult subjects. Two dose levels of the vaccine (2 μg LEP-F1 + 5 μg GLA-SE and 10 μg LEP-F1 + 5 μg GLA-SE) will be given by intramuscular administration on study Days 0, 28, and 56.

ELIGIBILITY:
Inclusion Criteria:

1. Males and females 18 years to 55 years of age.
2. Must be in good general health as confirmed by a medical history and physical exam.
3. Female subjects of childbearing potential must have a negative serum pregnancy test at screening and a negative urine pregnancy test on the day of each study vaccination, must not be breast-feeding, and are required to use one of the following methods of contraception from enrollment (Day 0) in study until 30 days after last injection (only if in sexual relationships with men): hormonal (e.g. oral, transdermal, intravaginal, implant, or injection); double barrier (i.e., condom, diaphragm, or cervical cap with spermicide); intrauterine device (IUD) or system (IUS); vasectomized partner (6 months minimum); or abstinence; bilateral tubal ligation (if no conception post-procedure); tubal occlusion; or bilateral salpingectomy. These precautions are necessary due to unknown effects that LEP-F1 + GLA-SE might cause in a fetus or newborn infant. Women are considered non-child-bearing potential if they are post-menopausal (defined as at least 12 months spontaneous amenorrhea and confirmed with FSH > 40 mIU/ml) or have had documented hysterectomy and/or oophorectomy.
4. The following screening laboratory values must be within the normal ranges or not clinically significant as determined by the Investigator and approved by the Medical Monitor: sodium, potassium, BUN, ALT, AST, total bilirubin, alkaline phosphatase, creatinine, fasting glucose, total WBC count, hemoglobin, and platelet count. Abnormal results may be repeated once for confirmation at Investigator discretion.
5. The following serology tests must be negative: HIV 1/2 antibody, hepatitis B surface antigen (HBsAg), QuantiFERON®-TB Gold (QFT), and hepatitis C virus (HCV) antibody.
6. Negative test for recreational drugs and alcohol per Clinical Research Unit standards.
7. Normal or not clinically significant urinalysis as determined by the study clinician or designee. Abnormal results may be repeated at Investigator discretion.
8. Must be capable of completing a study memory aid in English.
9. Must give informed consent, be able and willing to make all evaluation visits, be reachable by telephone or personal contact by the study site personnel, and have a permanent address.

Exclusion Criteria:

1. History of infection with M. leprae or previous exposure to M. leprae vaccines or experimental products containing GLA-SE.
2. History of BCG vaccination.
3. History of active or documented latent TB.
4. History of previous infection with other non-tuberculous mycobacteria.
5. Travel to or residence in India, Brazil, or Indonesia for more than 6 months.
6. Participation in another experimental protocol and/or receipt of any investigational products within the past 3 months prior to Screening.
7. Treatment with immunosuppressive drugs (e.g., oral or injected steroids, such as prednisone; high dose inhaled steroids) or cytotoxic therapies (e.g., chemotherapy drugs or radiation) in the past 6 months prior to Screening.
8. Received a blood transfusion within past 3 months prior to Screening.
9. Donated blood products (platelets, whole blood, plasma, etc.) within past one month prior to Screening.
10. Received any vaccine within past 1 month prior to Screening or have any planned immunizations while on study, with the exception of seasonal influenza vaccine which can be given after 1 month post the third study injection (Day 84).
11. History of autoimmune disease or other causes of immunosuppressive states.
12. History of any other acute or chronic illness (including cardiovascular, pulmonary, neurological, hepatic, rheumatic, hematological, metabolic or renal disorders, uncontrolled hypertension), or use of medication that, in the opinion of the Principal Investigator, may interfere with the evaluation of the safety or immunogenicity of the vaccine.
13. Rash, tattoos, or any other dermatological condition that could adversely affect the vaccine injection site or interfere with its evaluation.
14. BMI ≥ 32.
15. Hypertension (systolic > 150 or diastolic > 95) at screening and Day 0.
16. History of significant psychiatric illness with current use of medication.
17. Known or suspected alcohol or drug abuse within the past 6 months prior to Screening.
18. Chronic tobacco user (> 20 pack years).
19. Subjects with a history of previous anaphylaxis or severe allergic reaction to vaccines or unknown allergens.
20. Subjects who are unlikely to cooperate with the requirements of the study protocol.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 24 (Actual)
Dates: Start 2017-10-02 (Actual); Primary Completion 2019-03-05 (Actual); Study Completion 2019-03-05 (Actual)

PRIMARY OUTCOMES:
Number of adverse events | 421 days
  Solicited and unsolicited adverse events will be recorded for 28 days following each study injection; serious adverse events and adverse events of special interest will be recorded for the duration of the study.

SECONDARY OUTCOMES:
Immunogenicity (IgG antibody and T cell responses to LEP-F1) | Days 0, 35, and 63
  Immunogenicity will be evaluated by measuring humoral and cellular responses to LEP-F1 + GLA-SE at specified timepoints.

CONTACTS AND LOCATIONS:
Overall Officials: Corey Casper, MD, MPH, Study Director — Access to Advanced Health Institute (AAHI)
Locations (1):
- Covance Clinical Research Unit, Madison, Wisconsin, United States

IPD SHARING:
Plan to Share IPD: No